CLINICAL TRIAL: NCT02432820
Title: Assessment of 3D Transperineal Ultrasound Imaging With Matrix Array Transducers as a Potential Imaging Modality for Adaptive Prostate and Post-Prostatectomy Radiotherapy
Brief Title: Assessment of 3D Transperineal Ultrasound Imaging w/ Matrix Array Transducers in Prostate Radiotherapy
Status: Terminated | Type: Observational
Why Stopped: Business decision
Sponsor: Stanford University (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB-33012; PROS0070 (Other: OnCore)
Record Dates: First submitted 2015-04-16; First posted 2015-05-04 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
SPECIFIC STUDY AIMS

1. To evaluate congruence between pelvic anatomical structures segmented on MRI and/or CT scans co-registered with transperineal US scans acquired with an optically and/or electromagnetically tracked matrix array ultrasound transducer.
2. To estimate the achievable accuracy of anatomy tracking based on 3D US matrix-array transducer imaging and grey-level based image registration algorithms.

DETAILED DESCRIPTION:
SPECIFIC STUDY AIMS

1. To evaluate congruence between pelvic anatomical structures segmented on MRI and/or CT scans co-registered with transperineal US scans acquired with an optically and/or electromagnetically tracked matrix array ultrasound transducer.
2. To estimate the achievable accuracy of anatomy tracking based on 3D US matrix-array transducer imaging and grey-level based image registration algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Men that will undergo prostate radiotherapy as a primary treatment or post-prostatectomy.
* Age 18 or older
* Ability to understand and sign informed consent

Exclusion Criteria:

* Younger than 18 yrs old
* Inability to provide written and spoken consent.
* Patients with implanted actively controlled devices that may be subject to electromagnetic interference from the UroNav/PervuNav electromagnetic tracking used in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer patients being treated at Stanford Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in dose-volume histogram (DVH) indices in prostate images | 1 year
  The overall purpose of this study is to evaluate the ability of 3D ultrasound (US) to visualize the prostate with sufficient clarity and reliability to monitor and model anatomy motion and deformation. If this research study is successful in its findings, this mode of ultrasound imaging will have the ability to be adapted for the purposes of cost-efficient prostate radiotherapy.
Changes in dose-volume histogram (DVH) indices in bladder images | 1 year
  The overall purpose of this study is to evaluate the ability of 3D ultrasound (US) to visualize the bladder with sufficient clarity and reliability to monitor and model anatomy motion and deformation. If this research study is successful in its findings, this mode of ultrasound imaging will have the ability to be adapted for the purposes of cost-efficient prostate radiotherapy.
Changes in dose-volume histogram (DVH) indices in rectal wall images | 1 year
  The overall purpose of this study is to evaluate the ability of 3D ultrasound (US) to visualize the rectal wall with sufficient clarity and reliability to monitor and model anatomy motion and deformation. If this research study is successful in its findings, this mode of ultrasound imaging will have the ability to be adapted for the purposes of cost-efficient prostate radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitre Hristov, Principal Investigator — Stanford University; Steven Hancock, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States